CLINICAL TRIAL: NCT03445741
Title: Effects of Different Intensities and Durations of Aerobic Exercise Training and Detraining on Metabolic, Hormonal Responses and Abdominal Obesity in Women With Metabolic Syndrome.
Brief Title: Efficacy of Various Aerobic Exercises on Abdominal Obesity in Women With Metabolic Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Füsun Ardıç, Professor M.D., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015TPF037
Record Dates: First submitted 2018-02-11; First posted 2018-02-26 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Metabolic Syndrome
Keywords: Aerobic exercise; Metabolic syndrome; Pedometer
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Participants are assigned to three groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised treadmill group (%70 VO2 max) (Active Comparator): Supervised treadmill group (%70 VO2 max) (group 1): The participants were instructed walking exercise at their target heart rate, (% 70 of maximum oxygen consumption) on a treadmill in Sports Rehabilitation Unit of Pamukkale University.
  Interventions: Other: Supervised treadmill group (%70 VO2 max) (group 1)
- Supervised treadmill group (%50 VO2 max) (Experimental): Supervised treadmill group (%50 VO2 max) (group 2): The participants were instructed walking exercise at their target heart rate, (% 50 of maximum oxygen consumption) on a treadmill in Sports Rehabilitation Unit of Pamukkale University.
  Interventions: Other: Supervised treadmill group (%50 VO2 max) (group 2)
- ECE PEDO pedometer group (%50 VO2 max) (Experimental): ECE PEDO pedometer group (%50 VO2 max) (group 3): The participants were instructed walking with ECE PEDO which the number of steps taken in a minute corresponding to target HR at % 50 of maximum oxygen consumption were provided.
  Interventions: Device: ECE PEDO pedometer group (%50 VO2 max) (group 3)

INTERVENTIONS:
Other: Supervised treadmill group (%70 VO2 max) (group 1) — An exercise prescription was developed for each woman on the basis of the data acquired from the baseline treadmill exercise test. Target heart rate (HR) corresponding to values of 70% VO2max were determined by the submaximal treadmill test. The participants were instructed walking at their target HR on a treadmill in Sports Rehabilitation Unit of Pamukkale University. HR was monitored by a Polar HR monitor (Polar Beat, Port, Washington, NY). During 12 weeks, 3 days in a week and 20 minutes per day walking program was applied.
  Arms: Supervised treadmill group (%70 VO2 max)
Other: Supervised treadmill group (%50 VO2 max) (group 2) — An exercise prescription was developed for each woman on the basis of the data acquired from the baseline treadmill exercise test. Target heart rate (HR) corresponding to values of 50% VO2max were determined by the submaximal treadmill test. The participants were instructed walking at their target HR on a treadmill in Sports Rehabilitation Unit of Pamukkale University. HR was monitored by a Polar HR monitor (Polar Beat, Port, Washington, NY). During 12 weeks, 5 days in a week and 30 minutes per day walking program was applied.
  Arms: Supervised treadmill group (%50 VO2 max)
Device: ECE PEDO pedometer group (%50 VO2 max) (group 3) — Target heart rate (HR) corresponding to values of 50 % VO2max were determined by the submaximal treadmill test. The number of steps taken in a minute corresponding to target HR was determined by a criterion pedometer and group 3 was instructed walking in this step range recorded to ECE PEDO giving audible feedback. During 12 weeks, 5 days in a week and 30 minutes per day walking program was applied.
  Arms: ECE PEDO pedometer group (%50 VO2 max)

SUMMARY:
Objective: To show metabolic and hormonal responses and effects on abdominal obesity of aerobic exercise in different intensity and duration and detraining period in women with metabolic syndrome.

DETAILED DESCRIPTION:
Objective: To show metabolic and hormonal responses and effects on abdominal obesity of aerobic exercise in different intensity and duration and detraining period in women with metabolic syndrome.

Methods: Fifty-one women with metabolic syndrome were divided into three groups: 12 weekly sessions of high intensity supervised treadmill group, respectively, at % 70 of maximum oxygen consumption (group I, n=17), low intensity supervised treadmill group, respectively at % 50 of maximum oxygen consumption (group II, n=17) and walking at low intensity, respectively at % 50 of maximum oxygen consumption with ECEPEDO pedometer (group III, n=17). Target heart rate (HR) corresponding to values of 50-70 % VO2max were determined by the submaximal treadmill test. Group 1 and 2 were instructed walking at their target HR on a treadmill. The number of steps taken in a minute corresponding to target HR was determined by a criterion pedometer and group 3 was instructed walking in this step range recorded to ECE PEDO giving audible feedback. Participants were evaluated by weight, BMI, waist circumference (WC), blood sugar, LDL, HDL and triglyceride; viseral fat, trunk fat and waist circumference by bioelectrical impedance device (VIScan); ergospirometric VO2max at baseline, 12-week and 4-week detraining period.

ELIGIBILITY:
Inclusion Criteria:

* eligible participants who meet the criteria for inclusion were women with metabolic syndrome diagnosis according to National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) criteria and were 25-65 years old.
* Participants were well communicative, motivated and willing to participate in the study.

Exclusion Criteria:

* The exclusion criteria were presence of uncontrolled hypertension, type 2 diabetes mellitus, atherosclerotic heart disease, using drugs to affect thyroid, lipids metabolism and insulin sensitization, musculoskeletal or systemic diseases contradicting the exercise, a neurological or psychiatric disease affecting cooperation and cognitive function.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
*Change from baseline in abdominal viseral fat and trunk fat and measured by VIScan at week 12 and 4-week detraining period. | Week 12 and week 16
  BIA device ViScan, designed to estimate visceral adiposity and trunk fat percentage. A wireless 'electrode belt' is placed on the bare midriff of the subject in supine position. The belt then uses dual frequency bio impedance (6.25 and 50 kHz) to measure trunk and visceral fat resistance and transmit the readings via infrared to the base unit.
*Change from baseline in weight (kilograms) at week 12 and 4- week detraining period. | Week 12 and week 16
  Weight was measured with weight scale.
*Change from baseline in Epinephrine/Adrenaline parameter at week 12 and 4- week detraining period. | Week 12 and week 16
  Fasting blood samples were collected at morning hours before exercise testing. To perform adrenaline values, a sum of blood were stored at -80 C for later study.
*Change from baseline in noradrenaline parameter at week 12 and 4- week detraining period. | Week 12 and week 16
  Fasting blood samples were collected at morning hours before exercise testing. To perform noradrenaline values, a sum of blood were stored at -80 C for later study.
*Change from baseline in free fatty acide parameter at week 12 and 4- week detraining period. | Week 12 and week 16
  Fasting blood samples were collected at morning hours before exercise testing. To perform free fatty acide values, a sum of blood were stored at -80 C for later study.
*Change from baseline in oxyntomodulin parameter at week 12 and 4- week detraining period. | Week 12 and week 16
  Fasting blood samples were collected at morning hours before exercise testing. To perform oxyntomodulin values, a sum of blood were stored at -80 C for later study.
*Change from baseline in glycerol parameter at week 12 and 4- week detraining period. | Week 12 and week 16
  Fasting blood samples were collected at morning hours before exercise testing. To perform glycerol values, a sum of blood were stored at -80 C for later study.

IPD SHARING:
Plan to Share IPD: Undecided